CLINICAL TRIAL: NCT06892587
Title: Intervention Effects on Health Promoting Behaviors and Factors Influencing Long-Term Behavior Change
Acronym: HYP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6510
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Overweight (BMI > 25); Obese Patients
Keywords: sustainable health behaviors; virtual healthy eating program; eating behavior intervention
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Intervention Model Description: Single blinded randomized controlled trial, pilot study.
Who Masked: Participant
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy YOU Virtual behavioral Intervention (Experimental): An interactive, virtual intervention in a group setting focusing on adapting behaviors to sustain healthy improvements in dietary intake and physical activity.
  Interventions: Behavioral: An 8-week virtual group intervention designed to promote sustainable health behavior changes in participants
- Standard of Care Weight management intervention (Active Comparator): An 8 week standard of care intervention consisting of informational flyers that can be implemented in a self paced manner.
  Interventions: Behavioral: Standard of care Nutritional Information

INTERVENTIONS:
Behavioral: An 8-week virtual group intervention designed to promote sustainable health behavior changes in participants — The Healthy YOU Program is an 8-week virtual group intervention designed to help participants make lasting health behavior changes, focusing on diet and physical activity. Delivered via confidential Zoom sessions, it offers flexibility and support in a group setting. Participants engage in facilitated discussions, interactive activities, and expert guidance.
  Participants receive a structured curriculum with a printed workbook, covering evidence-based topics like nutrition, exercise, and well-being. Learning methods include:
  Weekly Newsletters: Provide health tips, resources, and reflections to support behavior change.
  Facilitated Group Discussions: Live sessions to share experiences, ask questions, and support each other.
  Applied Activities: Hands-on tasks like meal planning and goal-setting to build confidence.
  Demonstrations: Live sessions on healthy cooking, home exercises, and overcoming barriers.
  The program encourages goal setting, progress tracking, and self-regulation.
  Arms: Healthy YOU Virtual behavioral Intervention
Behavioral: Standard of care Nutritional Information — The standard of care will involve providing participants with 8 weeks of nutrition information through printed handouts. These handouts will be generic, similar to materials typically provided by healthcare providers or available on public-facing health/nutrition websites. While they will cover the same topics as the experimental group, the handouts will contain only basic, publicly available nutritional information and will not include guidance for application. These handouts are also included in the Healthy YOU curriculum as background material for weekly class preparation. Participants will be instructed to review and utilize the handout information in a self-paced manner over the 8-week period.
  Arms: Standard of Care Weight management intervention

SUMMARY:
This study aims to compare the 8-week virtual Healthy YOU Program with a standard care intervention that sends weekly nutrition and healthy living tips via email. It will evaluate short- and long-term changes in health behaviors, such as diet, physical activity, biomarkers, and body composition. The study also seeks to identify factors that help participants make lasting health changes and explore how lifestyle interventions can improve overall health. Findings may guide future programs and support non-weight-focused approaches to chronic disease management and healthcare policy.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65
* BMI between 25.00 and 40.00

Exclusion Criteria:

* Pregnancy or lactation
* Existing or previous eating disorders
* Use of a medically prescribed diet
* Weight loss or gain of 3 kg or more in the past 3 months
* Use of medications or supplements for weight or chronic disease management (withing the last 3 months)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Eating Behavior Inventory (EBI) | Baseline, 8 weeks and 3 months post intervention.
  The Eating Behavior Inventory (EBI) measures behaviors that help with weight management. It includes 26 items based on a survey of behavior treatment manuals, and focuses on behaviors linked to weight loss. Each item is rated on a 5-point scale, from "never" to "always." The EBI looks at both healthy behaviors (e.g., "I carefully watch the quantity of food I eat") and unhealthy behaviors (e.g., "I eat quickly compared to most people"). Negative behaviors are scored in reverse, so higher scores on the EBI indicate more behaviors that support weight loss. Scores range from 26 to 130.
Dietary Intake Patterns | Baseline, 8 weeks and 3 months post intervention.
  The ASA-24 Dietary Assessment Tool will be used to document foods and supplements consumed over a 3 day period (2 weekdays and a weekend day). Changes in sugar, sodium, and fat intake will be measured (with lower amounts indicating better outcomes) as well as changes in fruit and vegetable intake, fiber intake, and Healthy Eating Index score where higher amounts indicating better outcomes.
Physical Activity Levels | Baseline, 8 weeks and 3 months post intervention.
  Physical Activity levels measured by GODIN Physical Activity Assessment. Increases in frequency, time, type, and intensity of exercise would be associated with better outcomes.
Sustained Healthy Behaviors | 3 months post conclusion of intervention program.
  One or more diet or physical activity behaviors associated with a "better outcome" as measured by the ASA24 diet recall or the GODIN Physical Activity Assessment remains the same or better at the 3 month follow up mark as compared to baseline and post treatment visits.

SECONDARY OUTCOMES:
Total cholesterol | Baseline, 8 weeks and 3 months post intervention.
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
LDL Cholesterol | Baseline, 8 weeks and 3 months post intervention.
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
HDL Cholesterol | Baseline, 8 weeks and 3 months post intervention.
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Triglycerides | Baseline, 8 weeks and 3 months post intervention.
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
HemoglobinA 1c (HbA1c): Average blood sugar levels over 2-3 months. | Baseline, 8 weeks and 3 months post intervention.
  Measured with a point of care instrument that is a fully automated boronate affinity assay to determine the percentage of hemoglobin A1c in human whole blood.
Brachial Blood Pressure | Baseline, 8 weeks and 3 months post intervention.
  Measured with a point of care device that measures central (aortic) blood pressure and brachial blood pressure. It is based on a method called arterial tonometry.
Aortic Blood Pressure | Baseline, 8 weeks and 3 months post intervention.
  Measured with a point of care device that measures central (aortic) blood pressure and brachial blood pressure. It is based on a method called arterial tonometry.
Body Weight | Baseline, 8 weeks and 3 months post intervention.
  Measured using a standard stadiometer.
Body fat% | Baseline, 8 weeks and 3 months post intervention.
  Measured using Dual-Energy X-ray Absorptiometry (DEXA)
Lean Body Mass | Baseline, 8 weeks and 3 months post intervention.
  Measured using Dual-Energy X-ray Absorptiometry (DEXA).
Relationships Between Health Behaviors and Biomarkers/Body Composition | 8 weeks and 3 months post intervention.
  We'll assess any correlations between changes in health behaviors (dietary intake and physical activity) and improvements in biomarkers (e.g., cholesterol, blood pressure) and body composition (e.g., body fat percentage, muscle mass).
Self Efficacy | Baseline, 8 weeks and 3 months post intervention.
  A 10 item survey that assesses a person's overall self-confidence in their capacity to handle and overcome obstacles, perform tasks, and manage stress in different areas of life. Higher scores are associated with better outcomes.
Social Support | Baseline, 8 weeks and 3 months post intervention.
  A survey which measures how much support an individual feels they receive from their social network, including family, friends, and significant others. The scale evaluates the individual's perception of the availability, adequacy, and quality of social support in times of need. Higher scores are associated with better outcomes (higher social support).
Sleep quality | Baseline, 8 weeks and 3 months post intervention.
  Measured with the Pittsburgh Sleep Quality Index (PSQI). This survey contains 19 self-rated questions (items), and the responses are used to generate a total score. These items are divided into 7 components, each evaluating a different aspect of sleep quality. A total score of less than 5 suggests good sleep quality, with minimal sleep problems or disturbances. A total score of 5 or higher typically indicates poor sleep quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Food and Nutrition Clinical Research Lab, Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No